CLINICAL TRIAL: NCT02517281
Title: Prospective Clinical and Biologic Study of Secondary Cutaneous Effects in Targeted Cancer Therapies
Acronym: SKINTARGET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2010-A01052-37; 2010/1664 (Other: CSET number)
Record Dates: First submitted 2014-02-07; First posted 2015-08-07 (Estimated); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients having received targeted therapies (Experimental): Patients treated using targeted therapies
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy

SUMMARY:
The aim of the study is to do a descriptive analysis of the cutaneous toxicity observed in patients treated using targeted therapies in order to have a better understanding of the skin pathophysiology.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cancer beginning a targeted therapy
* Patients able to follow the protocol
* Age >/= 18 years old
* Signed inform consent

Exclusion Criteria:

* Patient unable to follow the protocol, having a non cooperative behavior or unable to come to follow up visits or unable to complete the study
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2011-07-12 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Number of clinical secondary effects bind to targeted therapies | Every 28 days up to 5 years
  Dermatological exam including questionnaire, clinical examination and photographies

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Robert, MD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Gustave Roussy Cancer Campus Grand Paris, Villejuif, Val De Marne, France